CLINICAL TRIAL: NCT04854746
Title: A Phase 1b, Multicenter, Randomized, Double-blind, Placebo-controlled Study to Determine the Safety and Immunogenicity of an Adenoviral-vector Based Oral Norovirus Vaccine Expressing GI.1 VP1 Administered Orally to Health Stable Older Adult Volunteers 55-80 Years of Age
Brief Title: Ph 1b: Safety & Immunogenicity of Ad5 Based Oral Norovirus Vaccine
Acronym: VXA-NVV-104
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vaxart (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: VXA-NVV-104
Record Dates: First submitted 2021-04-19; First posted 2021-04-22 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Norovirus Infections
Keywords: norovirus, oral vaccine, elderly
MeSH Terms: conditions — Caliciviridae Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1 Low Dose Active (Active Comparator): VXA-GI.1-NN tableted vaccine group, 2 doses (Day 1 and Day 29) at 1x10Log10
  Interventions: Biological: VXA-GI.1.NN
- Cohort 3 High Dose Active (Active Comparator): VXA-GI.1 tableted vaccine group, 2 doses (Day 1 and Day 29) at 1x10Log11
  Interventions: Biological: VXA-GI.1.NN
- Cohort 1 Low Dose Placebo (Placebo Comparator): Placebo tablets matching in number and appearance to active vaccine doses.
  Interventions: Biological: Placebo Tablet
- Cohort 3 High Dose Placebo (Placebo Comparator): Placebo tablets matching in number and appearance to active vaccine doses.
  Interventions: Biological: Placebo Tablet
- Cohort 2 Medium Dose Active (Active Comparator): VXA-GI.1 tableted vaccine group, 2 doses (Day 1 and Day 29) at 3x10Log10
  Interventions: Biological: VXA-GI.1.NN
- Cohort 2 Medium Dose Placebo (Placebo Comparator): Placebo tablets matching in number and appearance to active vaccine doses.
  Interventions: Biological: Placebo Tablet

INTERVENTIONS:
Biological: VXA-GI.1.NN — GI.1 oral vaccine tablet
  Arms: Cohort 1 Low Dose Active; Cohort 2 Medium Dose Active; Cohort 3 High Dose Active
Biological: Placebo Tablet — Tablets matching in number and appearance to active vaccine tablets
  Arms: Cohort 1 Low Dose Placebo; Cohort 2 Medium Dose Placebo; Cohort 3 High Dose Placebo

SUMMARY:
A Phase 1b, multicenter, randomized, double-blind, placebo-controlled study to determine the safety and immunogenicity of an adenoviral-vector based oral norovirus vaccine expressing GI.1 VP1 administered orally to healthy older adult volunteers 55-80 years of age. The study is designed to assess the safety, tolerability, immunogenicity, and efficacy of 3 dose levels of vaccine with a 2-dose vaccination schedule (4 weeks apart) in healthy older adults (55 to 80 years old)

DETAILED DESCRIPTION:
A Phase 1b, multicenter, randomized, double-blind, placebo-controlled study to determine the safety and immunogenicity of an adenoviral-vector based oral norovirus vaccine expressing GI.1 VP1 administered orally to healthy older adult volunteers 55-80 years of age. The study is designed to assess the safety, tolerability, immunogenicity, and efficacy of 3 dose levels of vaccine with a 2-dose vaccination schedule (4 weeks apart) in healthy older adults (55 to 80 years old).

Subjects will we randomized in the study utilizing an age and dose escalation schedule. A Safety Monitoring Committee will provide oversight of the trial throughout the duration of the study.

ELIGIBILITY:
Inclusion Criteria

To be eligible for this study, participants must meet all the following:

Age

1. 55 to 80 years old inclusive at the time of signing the Informed Consent Form (ICF).

   Type of Participants
2. In stable and good general health, without significant medical illness, based on medical history, physical examination and vital signs at screening
3. Safety laboratory values within the following range criteria at screening:

   1. Laboratory value of < grade 1 elevation from normal or decrease from normal with no clinical significance (NCS) for alkaline phosphatase (ALP), alanine aminotransferase (ALT), aspartate aminotransferase (AST), and bilirubin,
   2. Laboratory value of < grade 1 from normal with no NCS for:

      * decreased: albumin, magnesium, total protein and phosphorous
      * elevated: amylase, BUN, CPK and creatine and;
      * elevated or decreased: calcium, glucose, potassium and sodium;
4. Body mass index (BMI) between 17 and 35 kg/m2 at screening
5. Available for all planned visits and phone calls, and willing to complete all protocol- defined procedures and assessments (including ability and willingness to swallow multiple small enteric-coated tablets per study dose).

   Gender and Reproductive Considerations
6. Male or female participants Female participants must provide a negative pregnancy test at screening and baseline or be at least one year post-menopausal or surgically sterile. Female participants of childbearing potential must be willing to use a reliable oral, implantable, transdermal or injectable contraceptive for 30 days prior to and until 60 days post last study drug administration. The form of contraception must be approved by the Investigator Contraception use by men should be consistent with local regulations regarding the methods of contraception for participants in clinical studies.

   Informed Consent
7. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.

Exclusion Criteria

The participants must be excluded from participating in the study if they meet any of the following:

Medical Conditions

1. Presence of significant uncontrolled medical or psychiatric illness (acute or chronic) including institution of new medical/surgical treatment or significant dose alteration for uncontrolled symptoms or drug toxicity within 3 months of screening and reconfirmed at baseline
2. Cancer, or treatment for cancer treatment, within past 3 years (excluding basal cell carcinoma or squamous cell carcinoma)
3. Presence of immunosuppression or medical condition possibly associated with impaired immune responsiveness, including diabetes mellitus
4. History of irritable bowel disease or other inflammatory digestive or gastrointestinal condition that could affect the distribution/safety evaluation of an orally administered vaccine targeting the mucosa of the small intestine.

   Such conditions may include but are not limited to:
   1. Esophageal Motility Disorder
   2. Malignancy
   3. Malabsorption
   4. Pancreaticobiliary disorders
   5. Irritable bowel syndrome
   6. Inflammatory Bowel Disease
   7. Surgical Resection
   8. GERD
   9. Hiatal Hernia
   10. Peptic Ulcer (History of cholecystectomy is not exclusionary)
5. History of any form of angioedema
6. History of serious reactions to vaccination such as anaphylaxis, respiratory problems, hives or abdominal pain
7. Diagnosed bleeding disorder or significant bruising or bleeding difficulties that could make blood draws problematic
8. Any condition that resulted in the absence or removal of the spleen
9. Acute disease within 72 hours prior to vaccination defined as the presence of a moderate or severe illness (as determined by the Investigator through medical history and physical exam). (Assessment may be repeated during screening period.)
10. Presence of a fever ≥ 38oC measured orally at baseline (Assessment may be repeated during screening period)
11. Any significant hospitalization within the last year which in the opinion of the investigator or sponsor could interfere with study participation.
12. Any of the following history or conditions that may lead to higher risk of clotting events and/or thrombocytopenia:

    1. Family or personal history of bleeding or thrombosis
    2. History of heparin-related thrombotic events, and/or receiving heparin treatments
    3. History of autoimmune or inflammatory disease
    4. Presence of any of the following conditions known to increase risk of thrombosis within 6 months prior to screening:

       * Recent surgery other than removal/biopsy of cutaneous lesions
       * Immobility (confined to bed or wheelchair for 3 or more successive days)
       * Head trauma with loss of consciousness or documented brain injury
       * Receipt of anticoagulants for prophylaxis of thrombosis
       * Recent clinically significant infection
13. Any other condition that in the clinical judgment of the investigator would jeopardize the safety or rights of a participant taking in the study, would render the participant unable to comply with the protocol or would interfere with the evaluation of the study endpoints Diagnostic Assessments
14. Positive human immunodeficiency virus (HIV), Hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV) tests at the screening visit
15. Stool sample with occult blood at screening
16. Positive urine drug screen for drugs of abuse at screening (postive test for marijuana is not exclusionary; however concurrent use of marijuana during the study Active period through Day 57 is prohibited)
17. Positive breath or urine alcohol test at screening and baseline Prior/Concurrent Therapy
18. Receipt of a licensed vaccine (including any COVID-19 vaccines under Emergency Use Authorization) within 14 days prior to baseline vaccination or planned administration during the study active period (Day 57)
19. Use of antibiotics, proton pump inhibitors, H2 blockers or antacids within 7 days prior to study drug administration or planned use during the active study period (Day 57)
20. Use of medications known to affect the immune function (e.g., systemic corticosteroids and others) within 2 weeks before study drug administration or planned use during the active study period (Day 57)
21. Daily use of nonsteroidal anti-inflammatory drugs within 7 days prior to study drug administration or planned use during the active study period (Day 57)
22. Administration of any investigational vaccine, drug or device within 8 weeks preceding study drug administration, or planned use within the duration of the study Other Exclusions
23. Donation or use of blood or blood products within 30 days prior to study drug administration or planned donation during the active study period (Day 57)
24. History of drug, alcohol or chemical abuse within 1 year of screening
25. History of hypersensitivity or allergic reaction to any component of the investigational vaccine, including but not limited to fish gelatin

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-04-26 (Actual); Primary Completion 2022-01-04 (Actual); Study Completion 2022-01-04 (Actual)

PRIMARY OUTCOMES:
Rate of Solicited Adverse Events | Day 1 (Vaccination) to 7 days post vaccination
  Safety
Rate of Unsolicited Adverse Events | Day 1 (Vaccination) to 28 days post vaccination
  Safety

SECONDARY OUTCOMES:
VP1 specific IgA ASC | Day 1 (Vaccination) to 7 days post vaccination
  Immunogenicity
Norovirus GI.1 histo-blood group antigen GBGA blocking antibodies (BT50) | Day 1 (Vaccination) to 7 days post vaccination
  Immunogenicity
VP1 specific serum IgG | Day 1 (Vaccination) to 7 days post vaccination
  Immunogenicity

CONTACTS AND LOCATIONS:
Overall Officials: David Liebowitz, MD, PhD, Study Chair — Vaxart, Inc.
Locations (3):
- United States (3):
  - WCCT, Cypress, California
  - Benchmark Research, New Orleans, Louisiana
  - Benchmark Research, Austin, Texas

IPD SHARING:
Plan to Share IPD: No
Study results will be summarized and presented by treatment arm comparisons. Individual subject data will not be shared with other researchers.